CLINICAL TRIAL: NCT04582396
Title: A Pilot Study of Stellate Ganglion Blockade + Psychoeducation to Reduce Cardiac Anxiety and PTSD Symptoms in Cardiac Arrest Survivors
Brief Title: Stellate Ganglion Blockade to Reduce Cardiac Anxiety and PTSD Symptoms in Cardiac Arrest Survivors
Acronym: SGB-PsychoED
Status: Terminated | Phase: Not Applicable | Type: Interventional
Why Stopped: majority of the participants had exclusion criteria of anticoagulant use
Sponsor: Columbia University (Other)
Collaborators: National Institute on Aging (NIA) (NIH)
Responsible Party: Principal Investigator, Sachin Agarwal, Assistant Professor of Neurology, Department of Neurology, Columbia University
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: AAAS8305; 5P30AG064198-02 (NIH)
Record Dates: First submitted 2020-10-05; First posted 2020-10-09 (Actual); Results first posted 2024-07-31 (Actual); Last update posted 2024-07-31 (Actual); Status verified 2024-07

CONDITIONS: PTSD; Cardiac Arrest; Anxiety and Fear; Sleep Disturbance; Health Behavior
MeSH Terms: conditions — Stress Disorders, Post-Traumatic; Heart Arrest; Anxiety Disorders; Parasomnias; Health Behavior | interventions — Saline Solution

STUDY DESIGN:
Intervention Model Description: This is a pilot RCT to gain preliminary evidence regarding the acceptability, tolerability, safety, and efficacy of a combined intervention of Stellate Ganglion Blockade and psychoeducation vs sham-procedure and psychoeducation on trauma symptoms and health behaviors in patients exhibiting early PTSD symptoms after cardiac arrest.
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Masking Description: In addition to the unblinded coordinator, and due to the nature of the study treatment, the person performing the procedure cannot be blinded (i.e. the person performing the procedure needs to assess the effectiveness of the block objective physical signs and symptoms), but is encouraged not to disclose the allocation to the patient or outcome assessors either before or after the procedure.
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Stellate Ganglion Block + Psychoeducation (Experimental): For the active SGB arm, 7 to 8 mL of ropivacaine, 0.5%, will be injected around and into the site of the ganglion once before the hospital discharge. They will also receive a 30 minutes session of psychoeducation by a health professional with experience working with CA patients.
  Interventions: Procedure: stellate ganglion block injection; Behavioral: Psychoeducation
- Normal saline injection + Psychoeducation (Placebo Comparator): For the sham procedure, 1 to 2 mL of preservative-free normal saline will be injected into deep musculature in the neck. They will also receive a 30 minutes session of psychoeducation by a health professional with experience working with CA patients.
  Interventions: Procedure: Normal saline injection; Behavioral: Psychoeducation

INTERVENTIONS:
Procedure: stellate ganglion block injection — A stellate ganglion block (SGB) is an injection of local anesthetic (numbing medicine) to block the nerves located on either side of the voice box in the neck. It will be administered in an inpatient monitored setting.
  Other Names: SGB injection
  Arms: Stellate Ganglion Block + Psychoeducation
Procedure: Normal saline injection — An injection of normal saline will be injected into muscle on either side of the voice box in the neck. It will be administered in an inpatient monitored setting.
  Other Names: Sham procedure
  Arms: Normal saline injection + Psychoeducation
Behavioral: Psychoeducation — The session will be 30 minutes in duration, to be administered by a health professional with experience working with CA patients, the goal will be to establish rapport and help patient identify anxious situations, thoughts, and bodily feelings related their recent CA that could lead to avoidant behavior.
  Explain how many of these feelings are common in CA survivors, and they are often unrelated to their risk of its recurrence. Explain how the body has a fight-or-flight system that is controlled in part by the stellate ganglion and explain how blocking the action of this part of the body can reduce the feelings of anxiety that commonly occur. Discuss how certain activities such as exercise can increase feelings of anxiety around bodily sensations, but continued engagement could reduce that fear and that exercise is helpful for recovering from CA

SUMMARY:
This is a pilot randomized controlled trial (RCT) to gain preliminary evidence regarding the acceptability, tolerability, safety, and efficacy of a combined intervention of Stellate Ganglion Blockade (SGB) and psychoeducation on trauma symptoms and health behaviors in patients exhibiting early PTSD symptoms after cardiac arrest (CA).

Primary Aim 1 (Feasibility outcomes): Gain preliminary evidence regarding the acceptability, tolerability, and safety of conducting a randomized trial that evaluates a single SGB treatment in conjunction with psychoeducation among CA patients with early PTSD symptoms.

Secondary Aim 1 (Treatment-related outcomes): Test, whether SGB/psychoeducation treatment in CA patients with clinically significant PTSD symptoms is associated with reduced cardiac anxiety, PTSD symptoms, and improved health behaviors (physical activity and sleep duration), assessed objectively by a wrist-worn accelerometer for 4 weeks post-discharge.

DETAILED DESCRIPTION:
Every year in the U.S., 500,000 people experience sudden cardiac arrest (CA), caused by electrical disturbances across cardiac tissue, leading to marked arrhythmia that ultimately results in the heart ceasing to pump blood to the brain, lungs, and other organs. Due to advances in bundled post-arrest care, cardio-cerebral resuscitation, and effective cooling protocols, a substantial proportion of patients who receive guideline-based care (nearly 1 in 3 for out-of-hospital and ~50% for in-hospital CA) now survive this once universally fatal condition. While most survivors retain their cognitive function and physical independence, many grapple with CA's psychological consequences in the context of learning that they were "clinically dead."

In particular, many describe the CA experience as traumatic, and up to 1 in 3 CA survivors subsequently develop posttraumatic stress disorder (PTSD). Not only is PTSD common in CA patients, but there is evidence that PTSD after CA may influence health behaviors and prognosis.

Treatment of early PTSD and cardiac anxiety symptoms after CA requires timely intervention. Recent studies show that SGB is a safe and acceptable intervention for reducing PTSD symptoms in combat veterans. SGB treatment has never been tested to treat PTSD induced by acute medical events such as CA.

ELIGIBILITY:
Inclusion criteria

1. Age 18 years or older
2. Fluent in English or Spanish
3. A diagnosis of cardiac arrest (CA)
4. Admitted to the New York-Presbyterian Hospital
5. Elevated symptoms of psychological distress a. PCL-5 > 32 with a minimum of 2 weeks after cardiac arrest

Exclusion criteria

1. A prior SGB treatment
2. Severe brain injury defined as Cerebral Performance Category Score ≥3, and/or significant aphasia, dysarthria, or cognitive impairment precluding ability to complete study questionnaires as determined by interviewer
3. Terminal non-cardiovascular illness (life expectancy <1 year)
4. Severe mental illness requiring urgent psychiatric hospitalization
5. Alcohol or substance abuse that would impede ability to complete study
6. Unavailable for telephone and in-person follow-up
7. Allergy to amide local anesthetics (e.g., ropivacaine, bupivacaine)
8. Pre-existing Horner's syndrome
9. Pregnancy
10. Current anticoagulant use
11. History of a bleeding disorder
12. Infection or mass at injection site

Ages: 18 Years to 85 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 1 (Actual)
Dates: Start 2021-03-11 (Actual); Primary Completion 2021-04-19 (Actual); Study Completion 2021-04-19 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Sachin Agarwal, MD, MPH, Principal Investigator — Columbia University/New York Presbyterian; Ian M Kronish, MD, MPH, Study Director — Columbia University
Locations (1):
- Columbia University Medical Center/New York Presbyterian, New York, New York, United States

IPD SHARING:
Plan to Share IPD: Yes
De-identified data will be made available upon request to the study principal investigator.
Supporting Information: Study Protocol, SAP, ICF
Time Frame: Data will become available on August 1, 2021, and will be available until August 1, 2025.
Access Criteria: For whom: Researchers who provide a methodologically sound protocol. For what analyses: To achieve aims in the approved protocol.

RESULTS

PARTICIPANT FLOW:
Groups:
- Stellate Ganglion Block + Psychoeducation: For the active SGB arm, 7 to 8 mL of ropivacaine, 0.5%, will be injected around and into the site of the ganglion once before the hospital discharge. They will also receive a 30 minutes session of psychoeducation by a health professional with experience working with CA patients.
  stellate ganglion block injection: A stellate ganglion block (SGB) is an injection of local anesthetic (numbing medicine) to block the nerves located on either side of the voice box in the neck. It will be administered in an inpatient monitored setting.
  Psychoeducation: The session will be 30 minutes in duration, to be administered by a health professional with experience working with CA patients, the goal will be to establish rapport and help patient identify anxious situations, thoughts, and bodily feelings related their recent CA that could lead to avoidant behavior.
  Explain how many of these feelings are common in CA survivors, and they are often unrelated to their risk of its recurrence. Explain how the body has a fight-or-flight system that is controlled in part by the stellate ganglion and explain how blocking the action of this part of the body can reduce the feelings of anxiety that commonly occur. Discuss how certain activities such as exercise can increase feelings of anxiety around bodily sensations, but continued engagement could reduce that fear and that exercise is helpful for recovering from CA
- Normal Saline Injection + Psychoeducation: For the sham procedure, 1 to 2 mL of preservative-free normal saline will be injected into deep musculature in the neck. They will also receive a 30 minutes session of psychoeducation by a health professional with experience working with CA patients.
  Normal saline injection: An injection of normal saline will be injected into muscle on either side of the voice box in the neck. It will be administered in an inpatient monitored setting.
  Psychoeducation: The session will be 30 minutes in duration, to be administered by a health professional with experience working with CA patients, the goal will be to establish rapport and help patient identify anxious situations, thoughts, and bodily feelings related their recent CA that could lead to avoidant behavior.
  Explain how many of these feelings are common in CA survivors, and they are often unrelated to their risk of its recurrence. Explain how the body has a fight-or-flight system that is controlled in part by the stellate ganglion and explain how blocking the action of this part of the body can reduce the feelings of anxiety that commonly occur. Discuss how certain activities such as exercise can increase feelings of anxiety around bodily sensations, but continued engagement could reduce that fear and that exercise is helpful for recovering from CA
Period: Overall Study
Arm/Group | Stellate Ganglion Block + Psychoeducation | Normal Saline Injection + Psychoeducation
Started | 0 | 1
Completed | 0 | 1
Not Completed | 0 | 0

BASELINE CHARACTERISTICS:
Population: No accrued participants were randomized to the Stellate Ganglion Block + Psychoeducation Group
Groups:
- Total: Total of all reporting groups
Arm/Group | Stellate Ganglion Block + Psychoeducation | Normal Saline Injection + Psychoeducation | Total
Number analyzed (Participants) | 0 | 1 | 1
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years |  | 0 | 0
  Between 18 and 65 years |  | 1 | 1
  >=65 years |  | 0 | 0
Sex: Female, Male [Count of Participants; unit: Participants]
  Female |  | 0 | 0
  Male |  | 1 | 1
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino |  | 1 | 1
  Not Hispanic or Latino |  | 0 | 0
  Unknown or Not Reported |  | 0 | 0
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native |  | 0 | 0
  Asian |  | 0 | 0
  Native Hawaiian or Other Pacific Islander |  | 0 | 0
  Black or African American |  | 0 | 0
  White |  | 0 | 0
  More than one race |  | 0 | 0
  Unknown or Not Reported |  | 1 | 1
Region of Enrollment [Number; unit: participants]
  United States |  | 1 | 1
Posttraumatic Stress Disorder Scale [Number; unit: units on a scale] — This is a 20-item self-report measure that assesses symptoms of PTSD. Each item can be scored on a scale of 0-4, "Not at all" (0), "A little bit" (1), "Moderately" (2), "Quite a bit" (3), and "Extremely" (4) are the eligible responses. There are five clusters that are assessed: items 1-5, items 6-7, items 8-14, and items 15-20. Each of these sub-scores are summed to receive a score between 0-80; a higher score indicating a higher severity of PTSD symptoms. The cutoff score that is indicative of probable PTSD is 31-33.
  units on a scale |  | 43 | 43
Cardiac Anxiety Questionnaire [Number; unit: units on a scale] — This is an 18-item questionnaire that assesses anxiety through three divided sub-scales: fear (items 10, 11, 13-18), avoidance (items 2, 5, 7, 9, 12), and attention (items 1, 3, 4, 6, 8). Each item is scored via the 5-point Likert scale: "Never" (0), "Rarely" (1). "Sometimes" (2), "Often" (3), and "Always" (4). Item responses are summed to receive a score between 0-72. Higher reported scores indicate a greater heart-focused anxiety.
  units on a scale |  | 19 | 19
Generalized Anxiety Disorder Scale - 7 questions [Number; unit: units on a scale] — This is a 7-item scale that assesses the presence of generalized anxiety disorder. Responses can be given as "Not at all" (0), "Several days" (1), "More than half the days" (2), and "Nearly every day" (3). These scores can be summed to produce a score between 0 and 21. Scores between 0-4 indicate minimal anxiety, scores between 5-9 indicate mild anxiety, scores between 10-14 indicate moderate anxiety, and scores greater than 15 indicate severe anxiety.
  units on a scale |  | 11 | 11
Patient Health Questionnaire depression scale- 8 items [Number; unit: units on a scale] — This is an 8-item scale that assesses depression, with responses to each item being: "Not at all" (0), "Several days" (1), "More than half the days" (2), and "Nearly every day" (3). The sub-scores are summed to result in a score from 0-24. Higher scores indicate higher indication of depression. Scores that are reported as 10 or above are assessed to be showing symptoms of depression.
  units on a scale |  | 6 | 6

OUTCOME MEASURES:

1. Primary Outcome: Proportion of Eligible Subjects Who Get Enrolled in the Trial
Description: This is designed to measure the feasibility of successful enrollment.
Time Frame: Baseline (pre-procedure)
Population: During the enrollment period, 11 patients reported elevated PTSD and/or cardiac anxiety scores (an initial eligibility requirement for our study). Of these 11 patients, 10 were prescribed anticoagulants, rendering them ineligible for the study since one of the exclusion criteria is current anticoagulant use. One patient was enrolled and completed all study procedures.
Measure: Count of Participants; unit: Participants
Groups:
- Eligible Participants: For the sham procedure, 1 to 2 mL of preservative-free normal saline will be injected into deep musculature in the neck. They will also receive a 30 minutes session of psychoeducation by a health professional with experience working with CA patients.
  Normal saline injection: An injection of normal saline will be injected into muscle on either side of the voice box in the neck. It will be administered in an inpatient monitored setting.
  Psychoeducation: The session will be 30 minutes in duration, to be administered by a health professional with experience working with CA patients, the goal will be to establish rapport and help patient identify anxious situations, thoughts, and bodily feelings related their recent CA that could lead to avoidant behavior.
  Explain how many of these feelings are common in CA survivors, and they are often unrelated to their risk of its recurrence. Explain how the body has a fight-or-flight system that is controlled in part by the stellate ganglion and explain how blocking the action of this part of the body can reduce the feelings of anxiety that commonly occur. Discuss how certain activities such as exercise can increase feelings of anxiety around bodily sensations, but continued engagement could reduce that fear and that exercise is helpful for recovering from CA
Arm/Group | Eligible Participants
Number analyzed (Participants) | 11
Participants | 1

2. Primary Outcome: Number of Patients Recruited Per Month
Description: This is designed to measure the rate of enrollment, with <4 patients/month considered not meeting outcome
Time Frame: Assessed at 10 Month from the beginning of enrollment
Population: as for outcome 1
Measure: Count of Participants; unit: Participants
Arm/Group | Eligible Participants
Number analyzed (Participants) | 11
Participants | 1

3. Primary Outcome: Proportion of Participants Who Complete the 4-weeks Assessments
Description: This is designed to assess the short-term attrition and lost to follow-up up to 4 weeks post-enrollment.
Time Frame: 4 weeks post-enrollment
Population: There were no participants randomized to the Stellate Ganglion Block + Psychoeducation arm
Measure: Count of Participants; unit: Participants
Arm/Group | Eligible Participants
Number analyzed (Participants) | 1
Participants | 1

4. Primary Outcome: Proportion of Participants Who Complete the 12-weeks Assessments
Description: This is designed to assess the long-term attrition and lost to follow-up up to 12 weeks post-enrollment.
Time Frame: 12-weeks post-procedure
Population: There were no participants randomized to the Stellate Ganglion Block + Psychoeducation arm
Measure: Count of Participants; unit: Participants
Arm/Group | Eligible Participants
Number analyzed (Participants) | 1
Participants | 1

5. Primary Outcome: Horner's Syndrome
Description: Horner syndrome is a condition that affects the face and eye on one side of the body, being caused by a disrupted nerve pathway from the brain to the head and neck. This syndrome can be assessed through a visual exam, involving the observation of decreased pupil size, a drooping eyelid and decreased sweating on the affected side of the face.
Time Frame: Immediately post-procedure
Population: 11 patients reported elevated PTSD and/or cardiac anxiety scores (an initial eligibility requirement for our study). Of these 11 patients, 10 were prescribed anticoagulants, rendering them ineligible for our study since one of the exclusion criteria is current anticoagulant use. One patient was enrolled and completed all study procedures.
Measure: Count of Participants; unit: Participants
Arm/Group | Eligible Participants
Number analyzed (Participants) | 1
Participants | 1

6. Primary Outcome: Treatment Expectancy Eligibility Questionnaire
Description: This is a questionnaire that assesses the number of participants with credibility. Through this questionnaire, whether the participant will proceed through the study will be determined.
Time Frame: Immediately post-procedure
Population: 11 patients reported elevated PTSD and/or cardiac anxiety scores (an initial eligibility requirement for our study). Of these 11 patients, we learned that a majority (10 out of 11) were prescribed anticoagulants, rendering them ineligible for our study since one of the exclusion criteria is current anticoagulant use. One patient was enrolled and completed all study procedures.
Measure: Count of Participants; unit: Participants
Arm/Group | Eligible Participants
Number analyzed (Participants) | 1
Participants | 1

7. Primary Outcome: The Proportion of Participants Completing the Check-list of Various Components of Psychoeducation
Description: This is designed to assess the feasibility of administering psychoeducation, with >80% of the components in the checklist as a threshold for success.
Time Frame: Assessed at baseline post-procedure
Population: There were no participants randomized to the Stellate Ganglion Block + Psychoeducation arm
Measure: Count of Participants; unit: Participants
Arm/Group | Eligible Participants
Number analyzed (Participants) | 1
Participants | 1

8. Primary Outcome: Total Actigraph Wear Time
Description: the proportion of participants with >80% of the total actigraph wear time. It is designed to assess the acceptability of actigraphy
Time Frame: Assessed at 4-weeks post-procedure
Population: as for outcome 6
Measure: Count of Participants; unit: Participants
Arm/Group | Eligible Participants
Number analyzed (Participants) | 1
Participants | 1

9. Secondary Outcome: Number of Participants With Posttraumatic Stress Disorder Using Posttraumatic Stress Disorder (PCL-5)
Description: This is a 20-item self-report measure that assesses symptoms of PTSD. Each item can be scored on a scale of 0-4, "Not at all" (0), "A little bit" (1), "Moderately" (2), "Quite a bit" (3), and "Extremely" (4) are the eligible responses. There are five clusters that are assessed: items 1-5, items 6-7, items 8-14, and items 15-20. Each of these sub-scores are summed to receive a score between 0-80; a higher score indicating a higher severity of PTSD symptoms. The cutoff score that is indicative of probable PTSD is 31-33.
Time Frame: Assessed pre-procedure and then repeated at 4-weeks post-procedure
Population: There were no participants randomized to the Stellate Ganglion Block + Psychoeducation arm
Measure: Count of Participants; unit: Participants
Arm/Group | Eligible Participants
Number analyzed (Participants) | 1
Participants | 1

10. Secondary Outcome: The Proportion of Participants With Clinically Significant Symptoms of Cardiac Anxiety
Description: The effect of SGB-PsychoED intervention on cardiac anxiety will be assessed using cardiac anxiety questionnaire (CAQ).This is an 18-item questionnaire that assesses anxiety through three divided sub-scales: fear (items 10, 11, 13-18), avoidance (items 2, 5, 7, 9, 12), and attention (items 1, 3, 4, 6, 8). Each item is scored via the 5-point Likert scale: "Never" (0), "Rarely" (1). "Sometimes" (2), "Often" (3), and "Always" (4). Item responses are summed to receive a score between 0-72. Higher reported scores indicate a greater heart-focused anxiety.
Time Frame: Assessed pre-procedure and then repeated at 4-weeks post-procedure
Population: as for outcome 6
Measure: Count of Participants; unit: Participants
Arm/Group | Eligible Participants
Number analyzed (Participants) | 1
Participants | 1

11. Secondary Outcome: The Proportion of Participants With Clinically Significant Symptoms of Generalized Anxiety Disorder.
Description: The effect of the intervention on generalized anxiety disorder will be assessed using the generalized anxiety disorder scale-7 (GAD-7). This is a 7-item scale that assesses the presence of generalized anxiety disorder. Responses can be given as "Not at all" (0), "Several days" (1), "More than half the days" (2), and "Nearly every day" (3). These scores can be summed to produce a score between 0 and 21. Scores between 0-4 indicate minimal anxiety, scores between 5-9 indicate mild anxiety, scores between 10-14 indicate moderate anxiety, and scores greater than 15 indicate severe anxiety.
Time Frame: Assessed pre-procedure and then repeated at 4-weeks post-procedure
Population: as for outcome 6
Measure: Count of Participants; unit: Participants
Arm/Group | Eligible Participants
Number analyzed (Participants) | 1
Participants | 1

12. Secondary Outcome: The Proportion of Participants With Clinically Significant Symptoms of Depression.
Description: The effect of SGB-PsychoED intervention on depression will be assessed using the eight-item Patient Health Questionnaire depression scale (PHQ-8). This is an 8-item scale that assesses depression, with responses to each item being: "Not at all" (0), "Several days" (1), "More than half the days" (2), and "Nearly every day" (3). The sub-scores are summed to result in a score from 0-24. Higher scores indicate higher indication of depression. Scores that are reported as 10 or above are assessed to be showing symptoms of depression.
Time Frame: Assessed pre-procedure and then repeated at 4-weeks post-procedure
Population: as for outcome 6
Measure: Count of Participants; unit: Participants
Arm/Group | Eligible Participants
Number analyzed (Participants) | 1
Participants | 1

13. Secondary Outcome: The Proportion of Participants With Moderate to High Levels of Physical Activity.
Description: Effect of SGB-PsychoED intervention on mean minutes/day of physical activity as measured by the objective actigraphy data
Time Frame: Assessed at 4-weeks post-discharge
Population: as for outcome 6
Measure: Count of Participants; unit: Participants
Arm/Group | Eligible Participants
Number analyzed (Participants) | 1
Participants | 1

14. Secondary Outcome: The Proportion of Participants With Reduced Duration of Sleep.
Description: Effect of SGB-PsychoED intervention on mean hours/day of sleep as measured by the objective actigraphy data
Time Frame: Assessed at 4-weeks post-discharge
Population: as for outcome 6
Measure: Count of Participants; unit: Participants
Arm/Group | Eligible Participants
Number analyzed (Participants) | 1
Participants | 1

ADVERSE EVENTS:
Time Frame: Adverse Event Data were collected for 4 weeks after the intervention was administered
Description: Study personnel received alerts whenever a study participant was admitted to NYP Hospital/CUIMC
Arm/Group | Stellate Ganglion Block + Psychoeducation | Normal Saline Injection + Psychoeducation
All-Cause Mortality (participants affected / at risk) | 0/0 | 0/1
Serious Adverse Events (participants affected / at risk) | 0/0 | 0/1
Other Adverse Events (participants affected / at risk) | 0/0 | 1/1
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Stellate Ganglion Block + Psychoeducation (N=0) | Normal Saline Injection + Psychoeducation (N=1)
Emergency Room visit (Gastrointestinal disorders) | 0 | 1 (2) — Emergency Department visit unrelated to the study, satisfactorily resolved without an inpatient admission. The study team was not required to take any further action.

LIMITATIONS AND CAVEATS:
The study did not reach the target enrollment and therefore was inconclusive for treatment-related outcomes. This would need to be addressed in a future study in an outpatient setting because we learned that a majority of the inpatients were prescribed anticoagulants while in the hospital, which rendered them ineligible for the study.

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No

DOCUMENTS (2):
  • Study Protocol and Statistical Analysis Plan (2021-06-16): https://cdn.clinicaltrials.gov/large-docs/96/NCT04582396/Prot_SAP_000.pdf
  • Informed Consent Form (2021-10-14): https://cdn.clinicaltrials.gov/large-docs/96/NCT04582396/ICF_001.pdf